CLINICAL TRIAL: NCT04498078
Title: The Effects of Creatine Supplementation in Autism Spectrum Disorder: a Randomized Placebo-controlled Trial
Brief Title: Creatine Supplementation in Autism Spectrum Disorder
Acronym: CREATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABL-21-AUCR
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Creatine (Experimental): Twenty grams per day b.i.d.
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine monohydrate (20 g per day)

SUMMARY:
Autism Spectrum Disorder (ASD) is accompanied by reduced levels of total creatine in right temporal-parietal junction and other brain regions of interest, and addressing this deficit by exogenous administration of creatine may have beneficial effects on brain metabolism and disease-specific clinical symptoms in patients suffering from ASD.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 years and above
* Informed consent signed by a parent or legal guardian or legal representative
* Diagnostic and Statistical Manual of Mental Disorders-IV criteria for ASD.

Exclusion Criteria:

* Pregnant or nursing female patients
* Non-pharmacologic therapy
* Current diagnosis of other mental disorder

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Brain creatine change | Change from Baseline Brain Creatine Levels at 6 Months
  Monitor change in brain creatine levels by magnetic resonance imaging

SECONDARY OUTCOMES:
Brain N-acetylaspartate change | Change from Baseline Brain N-acetylaspartate Levels at 6 Months
  Monitor change in brain N-acetylaspartate levels by magnetic resonance imaging
Autism Treatment Evaluation Checklist (ATEC) score | Change from Baseline ATEC Scores at 6 Months
  Monitor changes in ASD severity

OTHER OUTCOMES:
Number of Participants With Potentially Clinically Relevant Laboratory Metabolic Abnormalities | Number of Participants With Potentially Clinically Relevant Laboratory Metabolic Abnormalities at 6-Month Follow-up
  Abnormal metabolic criterion values include fasting serum aspartate aminotransferase ≥ 40 U/L, fasting serum alanine aminotransferase ≥ 56 U/L, fasting serum gamma-glutamyl transferase ≥ 48 U/L
Maximal oxygen uptake change | Change from Baseline Cardiorespiratory Capacity at 6 Months
  Monitor changes in maximal oxygen uptake during an incremental exercise test on a treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Study Chair — Applied Bioenergetics Lab
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be provide via institutional online depository
Supporting Information: CSR
Time Frame: From January 2022 to December 2022
Access Criteria: Free access

REFERENCES:
- [Background] Edmondson DA, Xia P, McNally Keehn R, Dydak U, Keehn B. A Magnetic Resonance Spectroscopy Study of Superior Visual Search Abilities in Children with Autism Spectrum Disorder. Autism Res. 2020 Apr;13(4):550-562. doi: 10.1002/aur.2258. Epub 2020 Jan 7. PMID 31909886